CLINICAL TRIAL: NCT05001724
Title: A Randomized, Open-Label, Active-Controlled, Multi-Center Study to Compare Efficacy, Safety, and Tolerability of KN046 Combined With Lenvatinib Versus Docetaxel in Subjects With Non-Small Cell Lung Cancer After Failure of Anti-PD-(L)1 Agent
Brief Title: KN046 Plus Lenvatinib in Subject With Advanced Non-Small Cell Lung Cancer in the Failure of Anti-PD-(L)1 Agent
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Because the efficacy data did not meet expectations, the sponsor decided to terminate the study.
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KN046-302
Record Dates: First submitted 2021-07-16; First posted 2021-08-12 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — lenvatinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: KN046 plus Lenvatinib RP3D. (Experimental): Experimental arm: Cohort 1: KN046 5mg/kg every 3 weeks + lenvatinib RP3D every day until progressive disease or unacceptable toxicity.
  Interventions: Biological: KN046; Drug: Lenvatinib
- Docetaxel (Active Comparator): Active Comparator: docetaxel 75 mg/m² every 3 weeks until progressive disease or unacceptable toxicity.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: KN046 — KN046 is 5 milligram per kilogram, every 3 weeks.
  Arms: Cohort 1: KN046 plus Lenvatinib RP3D.
Drug: Lenvatinib — Lenvatinib is RP3D milligram per day, every day.
  Arms: Cohort 1: KN046 plus Lenvatinib RP3D.
Drug: Docetaxel — Docetaxel is 75 milligram per Square meter, every 3 weeks.
  Arms: Docetaxel

SUMMARY:
This is a phase 2/3, multicenter, randomized, open, positive-controlled study of patients with advanced non-small cell lung cancer whose disease has progressed after prior anti-PD-(L)1 therapy. Subjects should have documented progressive disease during prior treatment with first- or second-line PD-(L)1 and platinum-containing dual-agent chemotherapy.Subjects will be randomized to two treatment groups in a 1:1 ratio.

Treatment Group: KN046 5mg/kg Q3W + lenvatinib recommended for phase III dose (RP3D) every day.

Control group: Docetaxel 75mg/m2 Q3W .

ELIGIBILITY:
Inclusion criteria:

* Has a histologically confirmed or cytologically confirmed diagnosis of advanced NSCLC;
* Non-squamous non-small cell lung cancer, no EGFR mutation or ALK rearrangement or ROS1 fusion, no known RET fusion or MET14 exon jump mutation; Squamous non-small cell lung cancer with no known EGFR mutation or ALK rearrangement or ROS1 fusion /RET fusion /MET14 exon jump mutation;
* Has received prior systemic treatment with first- or second-line PD-(L)1 and platinum-containing dual-agent chemotherapy for their advanced NSCLC;
* Has measurable disease;
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status;
* Has adequate organ function;
* Has a life expectancy of at least 3 months;
* If female of childbearing potential, have a negative serum pregnancy test within 7 days prior to first trial treatment;
* If female of childbearing potential or a male subject with a partner with childbearing potential, be willing to use a highly effective method of contraception (with a failure rate of less than 1.0% per year) from first study treatment to 24 weeks after completion of the trial treatment.

Exclusion Criteria:

* Untreated active central nervous system metastasis or leptomeningeal metastasis;
* Is currently participating and receiving an investigational drug or has participated in a study of an investigational drug within 4 weeks or within 5 times of half-life (no less than 2 weeks), whichever is shorter prior to the first dose of trial treatment;
* Major surgery for any reason, except diagnostic biopsy, within 4 weeks of the first administration of trial treatment and/or if the subject has not fully recovered from the surgery within 4 weeks of the first administration of trial treatment;
* Curative radiation within 3 months of the first dose of trial treatment;
* Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of trial treatment (with the exception of subjects with adrenal insufficiency, who may continue corticosteroids at physiologic replacement doses, equivalent to < 10 mg prednisone daily, inhaled steroids and topical use of steroids);
* Vaccination within 28 days of the first administration of trial treatment, except for administration of inactivated vaccines;
* Has interstitial lung disease, or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management;
* History or current active autoimmune disease that might deteriorate when receiving an immunostimulatory agent;
* Previous malignant disease;
* History of uncontrolled intercurrent illness;
* Prior therapy with any antibody/drug targeting T cell coregulatory proteins;
* Has received treatment with lenvatinib or docetaxel or VEGFR-TKI;
* Known severe hypersensitivity reactions to antibody drug;
* Is pregnant or breastfeeding;
* Other medical conditions that at the discretion of investigator interfere with the requirements of the trial in terms of safety or efficacy evaluation, or treatment compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
DLT | 28 days or 21 days
  Dose limit toxicity (phase 2)
OS | up to 2 years
  Overall survival (OS) was defined as the time from randomization to death due to any cause (phase 3).
PFS | up to 2 years
  Progression-free survival (PFS) was defined as the time from randomization grouping to the first documented disease progression or death from any cause as evaluated by the investigator according to RECIST 1.1 criteria (phase 3).

SECONDARY OUTCOMES:
ORR | up to 2 years
  Objective response rate (ORR) based on the RECIST 1.1 by principal investigator
DCR | up to 2 years
  Disease control rate (DCR) based on the RECIST 1.1 by principal investigator
DOR | up to 2 years
  Duration of response (DOR) based on the RECIST 1.1 by principal investigator
CBR | up to 2 years
  Clinical benefit rate (CBR) based on the RECIST 1.1 by independent review committee
TTR | up to 2 years
  Time to response (TTR) based on the RECIST 1.1 by independent review committee

OTHER OUTCOMES:
Safety endpoint | up to 2 years
  Serious adverse events (SAE), changes and abnormal findings in laboratory test, vital sign and physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD,PhD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No